CLINICAL TRIAL: NCT03403829
Title: A Phase III Randomized Trial of Maintenance Chemotherapy in High-metastatic Risk Nasopharyngeal Carcinoma Patients of N3 Stage
Brief Title: Maintenance Chemotherapy in High-metastatic Risk Nasopharyngeal Carcinoma Patients of N3 Stage
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-NPC001
Record Dates: First submitted 2017-12-27; First posted 2018-01-19 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maintenance arm (Experimental): Gemcitabine maintenance treatment
  Interventions: Drug: Gemcitabine; Radiation: standard chemoradiotherapy
- control arm (Sham Comparator): observe and follow-up
  Interventions: Radiation: standard chemoradiotherapy

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine maintenance chemotherapy
  Other Names: standard chemoradiotherapy
  Arms: maintenance arm
Radiation: standard chemoradiotherapy — standard chemoradiotherapy

SUMMARY:
Up to now, IMRT has largely improved the local control of locally advanced nasopharyngeal carcinoma (NPC), leaves the distant metastasis as the main treatment failure modality of patients with bulky lymph nodes (especially N3 stage). Although concurrent chemoradiotherapy (CCRT) continues to stand as the standard treatment of these patients, the role of adjuvant chemotherapy remains controversial due to its relatively severe toxicities and inferior compliance. However, our retrospective study of 2D-RT and IMRT era had proved adjuvant chemotherapy played key role in N3 NPC patients in terms of reducing distant metastasis and improving overall survival. Maintenance chemotherapy of gemicitabine single drug is promising with adequate efficacy and moderate toxicities. So we aim to conduct "A Phase III Randomized Trial of Maintenance Chemotherapy in High-metastatic Risk Nasopharyngeal Carcinoma Patients of N3 Stage" to evaluate the effectiveness and compliance of gemicitabine as maintenance chemotherapy in N3 nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
We aim to conduct "A Phase III Randomized Trial of Maintenance Chemotherapy in High-metastatic Risk Nasopharyngeal Carcinoma Patients of N3 Stage" to evaluate the effectiveness and compliance of gemicitabine as maintenance chemotherapy in N3 nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* AJCC/UICC 8th edition N3 nasopharyngeal carcinoma
* Pathology: WHO II/II
* No prior anti-tumor treatment
* Age 18-60
* KPS≥70
* Adequate blood supply
* Informed consent obtained

Exclusion Criteria:

* Pathology: WHO I
* Pregnant
* Combined with other malignant tumor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Distant metastatic free survival | 5 year
  from enrollment to distant metastatis

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, M.D, Principal Investigator — Fudan University Shanghai cancer centre
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, Shanghai Municipality, China